CLINICAL TRIAL: NCT04914442
Title: Eosinophilic Cystitis Mimicking Urothelial Neoplasia: A Retrospective Study
Brief Title: Eosinophilic Cystitis Mimicking Urothelial Neoplasia
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, Laboratory manager, Al-Azhar University
Other Study IDs: AUH210501
Record Dates: First submitted 2021-06-03; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Urinary Bladder Diseases
MeSH Terms: conditions — Urinary Bladder Diseases | interventions — Microscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Microscopic examination — All the studies cases are microscopically examined using the ordinary stains (hematoxylin and eosin) then the eosinophilic infiltration are counted in 10 high power field manually

SUMMARY:
We explored the potential etiology, clinical and histopathology presentation of the eosinophilic cystitis cases, clinically mimicking urothelial neoplasia. Surgical procedure and clinical outcome also evaluated. T

DETAILED DESCRIPTION:
A pooled 22 patients diagnosed with eosinophilic cystitis on microscopic examination in our hospital during four years were retrospectively studied.We explored the potential etiology, clinical and histopathology presentation of the eosinophilic cystitis cases, clinically mimicking urothelial neoplasia. Surgical procedure and clinical outcome also evaluated. Transurethral resection of the lesions were performed and pathologically examined, we re-examined the studied cases and made a clinical correlation.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected urothelial neoplasia

Exclusion Criteria:

* Patients who did not complete the follow up period

Ages: 10 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients from Al-Azhar Hospital Urology outpatient and inpatient clinic during 4 years ftarting from January 2017
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Eosinophil cell count | 1 day
  Each tissue slide is retrieved and examined to count the eosinphils in the submucosa, positive cases revelaed more than 90% eosinophils of the whole inflammatory cells

CONTACTS AND LOCATIONS:
Overall Officials: Abdulkarim Hasan, Principal Investigator — Al-Azhar University

IPD SHARING:
Plan to Share IPD: Undecided